CLINICAL TRIAL: NCT03265314
Title: Alternatives For Girls (AFG) LeadHer
Brief Title: LeadHer, a Gender-specific Teen Pregnancy Prevention Curriculum for Girls 15-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alternatives For Girls (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Celia Thomas, Chief Operating Officer, Alternatives For Girls
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LeadHer
Record Dates: First submitted 2017-08-24; First posted 2017-08-29 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Teenage Pregnancy

STUDY DESIGN:
Intervention Model Description: Person-level random control trial. Participants randomly assigned to intervention (LeadHer) OR control (Sassy Science). Unit of analysis is individual (not groups/clusters). Baseline data collection is before randomization, in enrollment sessions, to prevent differential attrition post-randomization. Randomization via database developed for project. Evaluation Strategies (AFG's independent partner) developed an automated randomization method via random number generator. All randomized participants are tracked for study duration. In database, the button disappears once randomization occurs. The button is not active until consent/assent and all baseline measures are input to database. This randomization will occur after enrollment session, once enough participants for a cohort are enrolled. This helps prevent post-random sample loss. Randomization is electronic, via database, before first session. Once randomization occurs, AFG contacts enrolled girls about which their assigned program.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LeadHer (Experimental): The LeadHer curriculum is presented to the target population over a total of 30 hours. The program addresses the following adult preparation subjects: Healthy relationships, Adolescent development, Healthy life skills, Educational and career success. The LeadHer curriculum is also accompanied by a mobile application.
  Interventions: Behavioral: LeadHer
- Sassy Science (Placebo Comparator): The Sassy Science curriculum is presented to the target population over a total of 30 hours. The program addresses the following subjects: States of Matter, Math, Engineering, Chemistry, Arts and Crafts, Sweet Treats and Celebrations. The curriculum does not have a mobile application.
  Interventions: Behavioral: Sassy Science

INTERVENTIONS:
Behavioral: LeadHer — The 30-hour curriculum is delivered for five hours per week, either split over multiple after school sessions or one five-hour-long session conducted at AFG headquarters or a community-based partner site.
  Arms: LeadHer
Behavioral: Sassy Science — The 30-hour curriculum is delivered for five hours per week, either split over multiple after school sessions or one five-hour-long session conducted at AFG headquarters or a community-based partner site.
  Arms: Sassy Science

SUMMARY:
Alternatives For Girls (AFG) is offering LeadHer as a gender-specific teen pregnancy prevention curriculum to girls between the ages of 14-19 years old who live in Wayne County, MI. The curriculum seeks to demonstrate that girls who participate in LeadHer will show increased rates of avoidance of unprotected sex, will show increased use of birth control and reduced rates of pregnancy. LeadHer will run over a 6-session period covering topics designed to prevent teen pregnancy and develop girls into leaders. The sessions will be co-led by youth (Peer Educators).

DETAILED DESCRIPTION:
LeadHer is a 30-hour curriculum provided under rigorous evaluation, random assignment protocols and covering factual information related to sexual intercourse, including the risks of sex, sexually transmitted infections and use of birth control, along with the following adult preparation topics: Healthy relationships, Adolescent development, Healthy life skills, and Educational and career success.

The project is designed to run for five years; years 2 through 4 will involve providing the intervention curriculum to a total of 300 girls. There will be a control group, Sassy Science running in tandem with LeadHer for 300 girls. Groups will take place at the Alternatives For Girls facility as well as off-site within the community at local schools, primarily during after-school hours and community centers.

ELIGIBILITY:
Inclusion Criteria:

* Grade level: 8th grade through high school graduation; Race/ethnicity or tribe: As reflected in the Detroit, Wayne County, Michigan communities: African American, Latina, White, Mixed Races. At the time of the latest U.S. Census data, teens in Detroit were 81.9% African American, 9.7% Latino/a, 4.4% Caucasian, and 3.9% other races/ethnicities; Risk characteristics: Many will be at-risk by virtue of living within 200% of the federal poverty guidelines, doing poorly in local schools, being exposed to gang activities, and being sexually active; Other characteristics: living in Wayne County at the start of the study.

Exclusion Criteria:

* Target population participants who are already in another pregnancy prevention program.

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Female and female-identifying participants.
Enrollment: 508 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Avoidance of unprotected sex | Up to 12 months post the beginning of intervention.
  Participants will refrain from having sex or avoid sex without protection.
Use of birth control | Up to 12 months post the beginning of intervention.
  Participants decided to have sex, they will use birth control.
Presence of pregnancy | Up to 12 months post the beginning of intervention.
  Participants will get pregnant.

SECONDARY OUTCOMES:
Participants will report increased knowledge about Healthy Relationships | Up to 12 months post the beginning of intervention.
  Participants will report increased knowledge regarding ways to develop healthy relationships with parent/trusted adults and regarding dating violence. This will be collected via pre-tests and post-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Celia Thomas, MPA, Principal Investigator — Alternatives For Girls
Locations (1):
- Alternatives For Girls, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
None, N/A.